CLINICAL TRIAL: NCT06572657
Title: Comparison of the Effects of Aerobic Exercise and Computerized Cognitive Stimulation in Patients With Schizophrenia - A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Professor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İsmailK
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Exercise; Computerized Cognitive Stimulation
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cognitive stimulation group (Experimental): cognitive stimulation
  Interventions: Other: cognitive stimulation
- physical exercise group (Experimental): physical exercise
  Interventions: Other: physical exercise
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: cognitive stimulation — cognitive stimulation
  Arms: cognitive stimulation group
Other: physical exercise — physical exercise
  Arms: physical exercise group

SUMMARY:
Schizophrenia is a chronic mental disorder characterized by the occurrence of both positive symptoms, such as hallucinations and delusions, and negative symptoms, such as apathy and withdrawal, repetition of cognitive skills and disorganization. There are approximately 20 million people with schizophrenia worldwide and this number will continue to increase every year.

DETAILED DESCRIPTION:
The aim of this study was to compare the effects of computer-based cognitive stimulation and aerobic/strengthening exercises on symptom severity, cognition and depression in schizophrenia patients receiving community mental health center services.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with schizophrenia by a physician according to DSM-V criteria Patients treated at TRSM Individuals diagnosed with schizophrenia between the ages of 20-60

Exclusion Criteria:

* Those who did not give consent to participate in the study Patients with a diagnosis other than schizophrenia Pregnancy Patients with chronic metabolic diseases such as diabetes, heart problems and cancer

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale | 12 weeks
  MOCA is a short cognitive assessment method developed to detect particularly mild stages of cognitive impairment.
Frontal Assessment Battery | 12 weeks
  Frontal Assessment Battery consists of six subtests for assessing executive functions; the scale is scored from 0 to 18, with higher scores indicating better frontal functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No